## **Informed Consent Form (ICF)**

Official Title: The Effect of Tele-Nursing Service on Patients' Pain and Activity Level in Patients

Diagnosed With Fibromyalgia

Unique Protocol ID: NTK

NCT Number: [NCTXXXXXXXX]

Document Date: October 21, 2023 (IRB Approval Date)

Sponsor: Çankırı Karatekin University

Principal Investigator: Assist. Prof. Nedret Tekin Kaya

IRB Approval: Çankırı Karatekin University Scientific Research Ethics Committee, Approval No:

2023/09

Facility Location: Çankırı Karatekin University, Kırkevler Mahallesi, Kastamonu Caddesi, No:244

Uluyazı Kampüsü 18200 Merkez Cankırı, Turkey

## **Informed Consent Form**

Dear Participant,

This study is a scientific research project titled "The Effect of Tele-Nursing Service on Patients' Pain and Activity Level in Patients Diagnosed with Fibromyalgia" The results obtained based on the answers you provide within the scope of the research will contribute to determining the effect of tele-nursing services on the pain and activity levels of patients with fibromyalgia. Participation in this research is voluntary. No payment will be requested from you for participating in this research, nor will you receive any additional payment for your participation.

Participation in our study is voluntary. No fee will be charged for participating in this study, and no additional payment will be made to you for participating. You have the right to decline to participate in the study or to withdraw at any time after agreeing to participate. Withdrawing from the study will not negatively affect your treatment and care process. The answers you provide as part of the study will be kept confidential, and your name will not be disclosed in any way. Your answers will provide data for scientific research.

We appreciate your honest answers to the questions.

Consent to Participate in the Study

I have read all the explanations in the Informed Consent Form. The researchers named below have provided me with written and verbal explanations regarding the study mentioned above and its purpose. I have asked the researchers all the questions that came to mind, and I fully

understand all the written and verbal explanations provided to me. I agree to participate in the study voluntarily. I consent to the use of my medical information. I understand that if I do not agree to participate in the study, my treatment will be carried out without interruption or omission.

Participant

First Name Last Name

Date

Signature